CLINICAL TRIAL: NCT06892119
Title: Dose-reduced Generic Plerixafor Efficacy of Autologous Hematopoietic Stem Cell Transplantation in Patients with Lymphoma and Myeloma
Brief Title: Generic Plerixafor Efficacy of Autologous Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Cesar Homero Gutierrez-Aguirre, Principal Investigator, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HE19-00013
Record Dates: First submitted 2019-12-09; First posted 2025-03-24 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Lymphoma; Myeloma
MeSH Terms: conditions — Lymphoma; Neoplasms, Plasma Cell

STUDY DESIGN:
Intervention Model Description: Parallel study comparing placebo vs generic plerixafor
Who Masked: Participant
Masking Description: The patient receive a subcutaenous application (placbe vs generic plerixafor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Generic plerixafor (Active Comparator): Use a reduced-dose of generic plerixafor (0.12 mcg/Kg)
  Interventions: Drug: Celrixafor
- Placebo (Placebo Comparator): Use of a subcutaenous application of saline solution
  Interventions: Drug: Celrixafor

INTERVENTIONS:
Drug: Celrixafor — Use a reduced-dose of generic plerixafor

SUMMARY:
Generic plerixafor use at reduced-dose for mobilization on HSCT transplant

DETAILED DESCRIPTION:
The objective of this study is to demonstrate that the use of a low dose of the generic form of a drug called plerixafor is effective in increasing the amount of hematopoietic cells (stem cells) in your blood, which will then be collected for your transplant. Plerixafor is a very effective medicine that is already used for this purpose, however its high cost limits its use in all patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lymphoma or multiple myeloma who are candidates for autoHSCT
* Patients > 18 years old who signed our informed consent
* Normal CBC count (Hb > 10, WBC 4.0-11.00, plt > 100,000)

Exclusion Criteria:

* Patients with HIV, Hepatitis C, Hepatitis B diagnosis
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Post-RD plerixafor increase in CD34+/μL pre-count, final CD34+ cell yield and harvest | 1 year
  The objective of this study is to demonstrate that the use of a low dose of the generic form of plerixafor is effective in increasing the amount of hematopoietic cells (stem cells).

CONTACTS AND LOCATIONS:
Overall Officials: Olga G Cantú-Rodríguez, MD, Study Chair — Universidad Autónoma de Nuevo León
Locations (1):
- Universidad Autónoma de Nuevo León, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gutierrez-Aguirre CH, Alvarado-Navarro DM, Palomares-Leal A, Mejia-Jaramillo G, Salazar-Riojas R, Leon AG, Colunga-Pedraza PR, Sotomayor-Duque G, Jaime-Perez JC, Cantu-Rodriguez OG, Del Carmen Tarin-Arzaga L, Flores-Jimenez JA, Gomez-Almaguer D. Reduced-dose plerixafor as a mobilization strategy in autologous hematopoietic cell transplantation: a proof of concept study. Transfusion. 2019 Dec;59(12):3721-3726. doi: 10.1111/trf.15547. Epub 2019 Oct 16. PMID 31618456